CLINICAL TRIAL: NCT05556668
Title: Role of Biodegradable Polydioxanone Biliary Stents for the Percutaneous Treatment of Benign Biliary Strictures.
Brief Title: Percutaneous Biodegradable Biliary Stents for the Treatment of Benign Biliary Strictures.
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Eva Criado, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: CSPT_ECP_2020_600
Record Dates: First submitted 2022-09-06; First posted 2022-09-27 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Biliary Stricture; Biliary Tract Diseases; Bile Duct Stricture; Bile Duct Injury; Stents; Obstructive Jaundice
MeSH Terms: conditions — Biliary Tract Diseases; Jaundice, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous placement of biodegradable biliary stents — Benign biliary strictures treated with polydioxanone (PPDX) stents (Ella-DV biliary stent, ELLACS, Hradec Králové, Czech Republic). The stents are implanted using a percutaneous transhepatic cholangiography. Before stent implantation, balloon bilioplasty is be performed.

SUMMARY:
To assess safety and effectiveness in the long term of percutaneous insertion of Biodegradable (BD) Biliary Stents for the treatment of benign biliary strictures, in a single center experience.

DETAILED DESCRIPTION:
This is an observational study (retrospective analysis on a prospective database) of patients that have been implanted a biodegradable stent in the biliary tree to treat benign stenosis.

From march 2011 until May 2020, a prospective collection of clinical data has been conducted in patients with symptomatic benign biliary strictures treated biodegradable polydioxanone stents. A strict follow-up protocol has been carried out according to standard practice (at 2, 4, 6 months and every 6 months up to 5 years). Once the follow-up is completed, the collected data will be analyzed, assessing the long term effectiveness and safety, but also other variables related to stent implantation and impact on patient's quality of life.

A subgroup analysis of anastomotic biliary strictures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old attended in the interventional radiology department for the implantation of a biodegradable biliary stent (BBS: ELLA-CS, Hradec Kralove, Czech Republic), for each stenosis, by percutaneous technique.
* Written informed consent given

Exclusion Criteria:

* Patients under 18 years old
* Patients with post-liver transplant biliary strictures
* Patients for whom no post-intervention follow-up data are available
* Patients in whom malignancy is demonstrated as a cause of the stricture after stent placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with symptomatic benign biliary strictures from Parc Tauli University Hospital referral area and derived from other referring Hospitals treated in our center with a BBS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Stent Primary Patency | Time from stent implantation to new intervention due to restenosis or occlusion detected by clinical signs and symptoms and confirmed by blood-test disturbances and/or imaging tests), assessed up to 60 months
  Time until new intervention due to re-stenosis or occlusion (detected by clinical signs and symptoms and confirmed by blood-test disturbances and/or imaging tests)
Adverse Events | From stent implantation to completion of follow-up, up to 5 years
  Major and minor complications. The Clavien-Dindo classification will be used for grading the severity of complications.

SECONDARY OUTCOMES:
Technical Success | Immediate (during procedure)
  To correctly deploy a biodegradable stent using a percutaneous approach covering the stricture with a residual stenosis of less than 30% of the lumen, and correct flow of contrast through it into the intestinal lumen
Length of Hospital Stay | nights from admission to perform the stent implantation to discharge of the patient from the hospital, assessed up to 365 days
  number of days that patients spend in hospital to have the stent inserted, including a 24-48h control cholangiogram

CONTACTS AND LOCATIONS:
Overall Officials: Eva Criado-Paredes, MD, Principal Investigator — Corporació Universitaria Parc Tauli
Locations (1):
- Hospital Parc Tauli Sabadell, Sabadell, Spain